CLINICAL TRIAL: NCT06110104
Title: Effect of Retrowalking Program Versus Whole Body Vibration on Quadriceps Muscle Torque in Patients With Chronic Knee Osteoarthritis
Brief Title: Effect of Retrowalking Program Versus Whole Body Vibration in Patients With Chronic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marwa Gamal Abd El Ghany Fathalla (Other)
Responsible Party: Sponsor-Investigator, Marwa Gamal Abd El Ghany Fathalla, cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: knee osteoarthritis patients
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
Keywords: quadriceps torque,quadriceps endurance,balance,funcitional disability.
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: interventions; the first intervention: The Routine physiotherapy program comprises a combination of closed kinetic chain and open kinetic chain exercises, including straight leg raising, isometric quadriceps, isometric hip adduction, terminal knee extension, semi-squat, and leg press for 6 weeks.
  the other intervention : Retro-walking program is about 10 min of supervised retro walking training 3 days a week for 6 weeks at their comfortable walking speed . The participants will be instructed to gradually increase their walking time up to 30 min over the 6-week period.
  the last intervention is whole body vibration is 3 days per week for 6 weeks. During the training, the participants will perform static squat training barefoot on the platform with bent knees (30° and 60°). The distance between the feet was consistent with the shoulders. the duration time, sets and total time will be increased progressively over the 6-week.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Experimental): they recieve Routine physiotherapy program comprises a combination of closed kinetic chain and open kinetic chain exercises, including straight leg raising, isometric quadriceps, isometric hip adduction, terminal knee extension, semi-squat, and leg press for 6 weeks.
  Interventions: Other: routine physiotherapy program for knee osteoarthritis
- Retro-walking group (Experimental): they recieve routine physiotherapy and Retro-walking program which is about 10 min of supervised retro walking training 3 days a week for 6 weeks at their comfortable walking speed . The participants will be instructed to gradually increase their walking time up to 30 min over the 6-week period.
  Interventions: Other: routine physiotherapy program for knee osteoarthritis; Other: Retro-walking program
- whole body vibration group (Experimental): they recieve routine physiotherapy and whole body vibration which is 3 days per week for 6 weeks. During the training, the participants will perform static squat training barefoot on the platform with bent knees (30° and 60°). The distance between the feet was consistent with the shoulders. the duration time, sets and total time will be increased progressively over the 6-week.
  Interventions: Other: routine physiotherapy program for knee osteoarthritis; Other: whole body vibration training

INTERVENTIONS:
Other: routine physiotherapy program for knee osteoarthritis — The Routine physiotherapy program comprises a combination of closed kinetic chain and open kinetic chain exercises, including straight leg raising, isometric quadriceps, isometric hip adduction, terminal knee extension, semi-squat, and leg press for 6 weeks.
Other: Retro-walking program — Retro-walking program is about 10 min of supervised retro walking training 3 days a week for 6 weeks at their comfortable walking speed . The participants will be instructed to gradually increase their walking time up to 30 min over the 6-week period.
  Arms: Retro-walking group
Other: whole body vibration training — whole body vibration is 3 days per week for 6 weeks. During the training, the participants will perform static squat training barefoot on the platform with bent knees (30° and 60°). The distance between the feet was consistent with the shoulders. the duration time, sets and total time will be increased progressively over the 6-week.
  Arms: whole body vibration group

SUMMARY:
Osteoarthritis is one of the most common degenerative joint disease that affects approximately more than 300 million people worldwide

DETAILED DESCRIPTION:
this study compare the efficacy of Retro-walking program and whole body vibration on quadriceps muscle torque,endurance, Balance and knee functional disability in patients with chronic unilateral knee Osteoarthritis . it has three groups. first group recieves The Routine physiotherapy program comprises a combination of closed kinetic chain and open kinetic chain exercises cause the least intraarticular inflammation, bone destruction, and pressure over the joint. the seconed group recieves routine physiotherapy and Retro-walking which is considered a safe Closed Kinematic Chain exercise since the compressive forces at the patello-femoral joint are reduced. it include improvement in muscle activation pattern, Reduction in adductor moment at knee during stance phase of gait and augmented stretch of hamstring muscle groups during the stride; all of these may have helped in reducing disability thus leading to improved function.It reduces quadriceps eccentric function, while the isometric and concentric quadriceps strength are preserved improved pain relief and aerobic fitness level, without aggravating symptoms following walking programs in patients with knee OA. the third group recieves routine physiotherapy program and Whole-body vibration training which is now a day's got its wider importance, especially in clinical cases. It has a role in maintaining balance, proprioception, blood circulation, and hormone level that enhances the effect on the neuromuscular system . it is a new type of exercise therapy, which mainly improves muscle coordination to optimize joint function .it is performed as a neuromuscular modality in muscle strength training . As it is safe, effective and potentially feasible treatment, WBV training has also been proposed for several musculoskeletal system diseases.

the study ethical committee number is NO:P.T.REC/012/004280. the total sample size are 45 (for 3 groups), 45 patients (15 patients per group).

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects are required to have a radiograph of the knee joints within 2 weeks of testing.

  2.Weight-bearing, fixed flexion radiographs of the knee were taken in the AP views .

  3.Radiographic evidence of knee OA.according to Kellgren and Lawrence classification scale (gradeIII) as 0,Normal and 4,Sever.

  4.Particepants age are 40-55 . 5.Knee pain for at least 3 month , with pain presenting at least 3 days a week during last month.

  6.functional limitations (patients with pain &stiffnes), The Arabic version of the western womac (ArWOMAC) scores (average 37) 7.ability to ambulate independently for at least 10 meters. 8.Ability to follow simple structures.

Exclusion Criteria:

* 1.(BMI) more ≥ 30. 2.History of knee surgery to knee within past 3 months 3.A systemic arthritic condition. 4.Any other muscular, joint or neurological condition affecting lower limb function.

  5.Physical therapy or an intra-articular injection in the knee within the past 3 months.

  6.Change in pain medications in the previous month. 7.Healthy participants, impairment conditions unrelated to gait conditions such as cardio- and respiratory-related diseases, people with lower limb amputations, and lower prosthetic limbs.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The estrogen via estrogen receptor mediates osteoarthritis cartilage degradation and accelerates the progression of cartilage loss increase disease risk in females more than males.
Enrollment: 45 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
quadriceps torque | 6 weeks
  hand-held dynamometer offers a reliable and valid method to quantify quadriceps strength in a clinical environmen .quadriceps peak torque obtained with an HHD is valid compared to an isokinetic dynamometer. it offers a less expensive and time-consuming way to obtain measures in a clinical environment. The torque peak (Nm) of the quadriceps will be measured by multiplying the force, acceleration of gravity and lever arm: [force (kg) × 9.81 × lever arm (m)]. Quadriceps torque (Nm) data were normalized by the body mass (kg) of each participant: torque (Nm)/body mass (kg).
quadriceps endurance | 6 weeks
  Fatigue resistance test assesses Quadriceps isometric endurance .The individuals will sit on a chair with their back straight and their hips and knees flexed at 90 degrees. A 5 kg weight will be secured with tape above the ankle (testing side), and leg alignment In relation to the horizontal plane measured by digital inclinometer.A stopwatch will use to record the time. The duration of time spent in this position is used to determine their knee extensor endurance capacity. If the knee extension position shifted at least five degrees from the horizontal plane , or the participant could not sustain the test leg in a horizontal position due to pain or fatigue, the test will be terminated.This Endurance testing protocol will be repeated three times, and the best effort will be taken for analysis. There is a rest period of three minutes between each testing trial. The same investigator will record the individuals' readings.
balance | 6 weeks
  Balance in knee osteoarthritis will be measured by Time up and go test During the test, all participants were asked to stand up from a chair without armrests and with a seat height of 44 cm, walk at a comfortable pace to a line 3 m away, cross the line and turn through 180°, walk back, and sit in their starting position. The use of an assistive device was allowed for those using one, but no verbal encouragement or personal assistance was given. After one pilot test, the average time of the two successive trials was recorded using a timer with an accuracy of 1/100 s.
knee functional disability | 6 weeks
  Functional disability will be assessed using the Arabic version of the Western Ontario and McMaster Universities Osteoarthritis index.
  The pain subscale includes five questions about pain .The stiffness subscale includes two questions about stiffness . The physical function subscale includes 17 questions about the degree of difficulty .Each of the 24 questions is graded either on a five-point Likert scale (0 to 4) or a 100 mm visual analogue scale (VAS)9ranging from 0 (no pain) to 100 (extreme pain).

CONTACTS AND LOCATIONS:
Overall Officials: manal mo ismail, PHD, Study Chair — Cairo University; sara mo samir, MSc, Study Director — Cairo University; Ahmed om abd el naem, MSc, Study Director — faculty of physical therapy cairouniversity; marwa ga amr, BSc, Principal Investigator — faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt